CLINICAL TRIAL: NCT00704691
Title: Open-Label, One Arm Pilot Investigation of Lenalidomide Therapy for Patients With Relapsed and/or Refractory, Peripheral T-Cell Lymphomas
Brief Title: Lenalidomide Therapy for Patients With Relapsed and/or Refractory, Peripheral T-Cell Lymphomas
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Closed due to futility with only 1 patient accrued
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F071108004; UAB 0663 (Other: Cancer Center department study number)
Record Dates: First submitted 2008-06-21; First posted 2008-06-25 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Peripheral T-cell Lymphomas; Adult T-cell Leukemia; Adult T-cell Lymphoma; Peripheral T-cell Lymphoma Unspecified; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large Cell Lymphoma; T/Null Cell Systemic Type; Cutaneous t-Cell Lymphoma With Nodal/Visceral Disease
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Leukemia-Lymphoma, Adult T-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide 25 mg as a daily oral dose days 1-21 followed by a 7 day rest period (28 day cycle) for 1-6 cycles

SUMMARY:
The purpose of this study is to:

* assess the effectiveness of lenalidomide for the treatment of patients with relapsed and or refractory peripheral T-cell lymphomas; and,
* assess the safety of lenalidomide.

There are reports suggesting a therapeutic benefit of thalidomide in patients with refractory and/or relapsed Non-Hodgkin's Lymphoma's (NHL) which have led to the formal investigation of lenalidomide in the treatment of relapsed NHL's.

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCL's) represent a subgroup of Non-Hodgkin's lymphomas with poor prognostic features. Compared to aggressive B-cell lymphomas, PTCL's often present with more advanced disease and sustain less durable remissions following treatment with chemotherapy. With standard anthracycline-based regimens such as CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone), PTCLs achieve inferior 5-year overall survival rates of around 40% compared to aggressive B-cell lymphomas whose 5-year overall survival rates reach 50-60%. While several salvage regimens have been established for B-cell lymphomas with moderate success, the guidelines for patients with relapsed and/or refractory PTCL's are less clear. Several reports suggest that the immunomodulatory drugs (IMiDs®) have clinical activity in this setting. The aim of this phase 2 study is to evaluate the activity of lenalidomide in relapsed and/or refractory PTCL's.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age 19 and over at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Patients with a confirmed diagnosis of peripheral T-cell lymphomas according to the World Health Organization (WHO) classification in the relapsed and/or refractory setting following prior anthracycline therapy. Subtypes of peripheral T-cell lymphomas which meet this criteria will include the following: adult T-cell leukemia/lymphoma, peripheral T-cell lymphoma unspecified, angioimmunoblastic T-cell lymphoma, anaplastic large-cell lymphoma, T/null cell, primary systemic type, subcutaneous panniculitis-like T-cell lymphoma, hepatosplenic gamma-delta T-cell lymphoma, and enteropathy-type T-cell lymphoma [33].
5. Patients with a history of PTCL or cutaneous T-cell lymphoma (CTCL) with nodal/visceral disease in the relapsed and/or refractory setting following prior anthracycline therapy. This includes ≥ 3-6 cycles of CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone) or an equivalent, CHOP-like regimen +/- radiation therapy. The definition for relapsed and refractory disease is provided in Appendix 5.
6. All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
7. At least one measurable lesion according to the International Working Group response criteria for non-Hodgkin's lymphoma (see Appendix 5).
8. ECOG performance status of less than or equal to 2 at study entry (see Appendix 2).
9. Laboratory test results within these ranges:

   * Absolute neutrophil count greater than or equal to 1.5 x 109/L
   * Platelet count greater than or equal to 100 x 109/L (>70 x 10^9/L if bone marrow was involved)
   * Serum creatinine less than or equal to 2.0 mg/dL
   * Total bilirubin less than or equal to 1.5 mg/dL
   * AST (SGOT) and ALT (SGPT) less than or equal to 2 x upper limit of normal (ULN) or less than or equal to 5 x ULN if hepatic metastases are present.
10. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to therapy and again within 24 hours of prescribing lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex* condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix 1: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

    * For patients who have latex allergies or whose partner(s) have latex allergies alternatives will be discussed.
11. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
12. Disease free of prior malignancies for greater than or equal to 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast
13. Able to take aspirin (81 mg) daily as prophylactic anticoagulation, if deemed necessary by investigator (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodorum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or treatments within the past 28 days.
9. Known positive for HIV or infectious hepatitis, type A, B or C.
10. (Other) Precursor T-cell lymphomas (including immature T-cell lymphomas/leukemias) and cutaneous T-cell lymphomas (CTCL) with skin as the only organ of involvement
11. Patients with prolonged QT interval on baseline EKG (>430 ms)
12. Equal to greater than grade 3 peripheral neuropathy.
13. Natural Killer (NK) cell lymphomas

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Response Rate to lenalidomide (CR,PR and unconfirmed complete responses | Efficacy assessments every 8 weeks with a final assessment performed at the end of Cycle 6 (wk 24).

SECONDARY OUTCOMES:
Toxicity of lenalidomide | Progressive disease during cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: James Foran, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States